CLINICAL TRIAL: NCT05518539
Title: Evaluation of Quality of Vision and Visual Outcomes With Bilateral Implantation of the Clareon PanOptix Intraocular Lens
Status: Completed | Type: Observational
Sponsor: Newsom Eye & Laser Center (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: THN-22-001
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Results first posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- The Clareon™ PanOptix™ Trifocal (toric and non-toric models): Bilateral implantation with the Clareon PanOptix Trifocal (toric and non-toric models)
  Interventions: Device: The Clareon™ PanOptix™ Trifocal (toric and non-toric models)

INTERVENTIONS:
Device: The Clareon™ PanOptix™ Trifocal (toric and non-toric models) — Bilateral implantation with the Clareon PanOptix Trifocal (toric and non-toric models)

SUMMARY:
To evaluate visual outcomes and quality of vision following bilateral implantation of the Clareon PanOptix intraocular lens (IOL) targeted for emmetropia.

DETAILED DESCRIPTION:
This study is a single-arm unmasked clinical evaluation study of binocular distance-corrected near (40 cm) visual acuity after successful bilateral cataract surgery. Subjects will be assessed pre-operatively, operatively and at 1 day, 1 month and 3 months post-operatively. Clinical evaluations will include administration of a visual disturbance questionnaire (QUVID), and a satisfaction questionnaire (IOLSAT), as well as measurement of bilateral visual acuity and manifest refraction.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in both eyes.

* Presenting for uncomplicated bilateral cataract surgery and have an interest in spectacle independence using a trifocal IOL
* Meet the requirements for on-label implantation of the trifocal IOL
* Gender: Males and Females.
* Age: 40 or older.
* Willing and able to provide written informed consent for participation in the study.
* Willing and able to comply with scheduled visits and other study procedures.
* Have good ocular health, with no pathology that compromises visual acuity (outside of residual refractive error and cataract).
* Expected visual potential of 20/25 Snellen (0.10 logMAR) or better in each eye.
* All eyes will be in the range of availability for Clareon PanOptix IOL and Clareon PanOptix Toric IOL. For cylinder below the Toric IOL indication (T3), an LRI will be used during surgery.

Exclusion Criteria:

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Patients with any corneal pathology (including corneal dystrophies, scaring, severe dry eye syndrome, irregular astigmatism, HOA) limiting or affecting visual potential.
* Patients with previous corneal refractive surgery.
* Patients with pre-existing ocular pathology, including maculopathy, ARMD, ERM, prior RD, and glaucoma limiting or affecting visual potential.
* Subjects who have an unstable acute or chronic disease or illness that would confound the results of this investigation (e.g., immunocompromised, connective tissue disease, clinically significant atopic disease, diabetes, and any other such disease or illness), that are known to affect postoperative visual acuity.
* Participation in any investigational drug or device trial within the previous 30 days prior to the start date of this trial (or currently participating).

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be presenting for cataract surgery who are interested in a reduced dependence on spectacles for near, intermediate and distance vision, and who are considered appropriate candidates for trifocal lens implantation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Newsom, MD, Principal Investigator — Newsom Eye & Laser Center
Locations (1):
- Newsom Eye & Laser Center, Sebring, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | The Clareon™ PanOptix™ Trifocal (Toric and Non-toric Models)
Started | 30
Completed | 24
Not Completed | 6
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | The Clareon™ PanOptix™ Trifocal (Toric and Non-toric Models)
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Binocular Distance-corrected Near (40 cm) Visual Acuity
Time Frame: 1 month postoperatively
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | The Clareon™ PanOptix™ Trifocal (Toric and Non-toric Models)
Number analyzed (Participants) | 24
logMAR | 0.00 (00.06)

2. Primary Outcome: Binocular Distance-corrected Near (40 cm) Visual Acuity
Time Frame: 3 months postoperatively
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | The Clareon™ PanOptix™ Trifocal (Toric and Non-toric Models)
Number analyzed (Participants) | 24
logMAR | 0.01 (0.10)

3. Secondary Outcome: Binocular Uncorrected Distance (6 m) Visual Acuity
Time Frame: 1 and 3 months postoperative
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | The Clareon™ PanOptix™ Trifocal (Toric and Non-toric Models)
Number analyzed (Participants) | 24
logMAR
  1 Month | 0.00 (0.08)
  3 Months | 0.02 (0.19)

4. Secondary Outcome: Binocular Uncorrected Intermediate (60 cm) Visual Acuity
Time Frame: 1 and 3 months postoperative
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | The Clareon™ PanOptix™ Trifocal (Toric and Non-toric Models)
Number analyzed (Participants) | 24
logMAR
  1 Month | -0.04 (0.08)
  3 Months | -0.08 (0.09)

5. Secondary Outcome: Binocular Uncorrected Near (40 cm) Visual Acuity
Time Frame: 1 and 3 months postoperative
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | The Clareon™ PanOptix™ Trifocal (Toric and Non-toric Models)
Number analyzed (Participants) | 24
logMAR
  1 Month | 0.04 (0.09)
  3 Months | 0.04 (0.12)

6. Secondary Outcome: Binocular Corrected Corrected Distance (6 m) Visual Acuity
Time Frame: 1 and 3 months postoperative
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | The Clareon™ PanOptix™ Trifocal (Toric and Non-toric Models)
Number analyzed (Participants) | 24
logMAR
  1 Month | -0.02 (0.07)
  3 Months | -0.04 (0.08)

7. Secondary Outcome: Binocular Distance-corrected Intermediate (60 cm) Visual Acuity
Time Frame: 1 and 3 months postoperative
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | The Clareon™ PanOptix™ Trifocal (Toric and Non-toric Models)
Number analyzed (Participants) | 24
logMAR
  1 Month | -0.04 (0.08)
  3 Months | -0.08 (0.10)

8. Secondary Outcome: Manifest Refraction
Description: spherical equivalent refraction and astigmatism less than or equal to 0.5 D.
Time Frame: 3 months postoperative
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | The Clareon™ PanOptix™ Trifocal (Toric and Non-toric Models)
Number analyzed (Participants) | 24
Number analyzed (eyes) | 48
eyes
  Manifest Refraction Spherical Equivalent | 46
  Astigmatism | 46

9. Secondary Outcome: Satisfaction Questionnaire
Description: The Intraocular Lens Satisfaction questionnaire (IOLSAT). Subjects were asked how often they needed to wear eyeglasses to see at distance, intermediate, and near. The percentage was calculated as (# of subjects responding "Never" or "Rarely") divided by (# of subjects) times 100. A higher percentage is a better outcome.
Time Frame: 3 months postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | The Clareon™ PanOptix™ Trifocal (Toric and Non-toric Models)
Number analyzed (Participants) | 24
Participants
  Spectacle independence distance (overall) | 24
  Spectacle independence intermediate (overall) | 22
  Spectacle independence near (overall) | 17

10. Secondary Outcome: Visual Disturbances Questionnaire
Description: Questionnaire for Visual Disturbances (QUVID).
Time Frame: 3 months postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | The Clareon™ PanOptix™ Trifocal (Toric and Non-toric Models)
Number analyzed (Participants) | 24
Participants
  Bothered quite a bit" or "Bothered very much" by starbursts | 3
  Bothered quite a bit" or "Bothered very much" by halos | 2
  Bothered quite a bit" or "Bothered very much" by glare | 0
  Bothered quite a bit" or "Bothered very much" by haze | 0
  Bothered quite a bit" or "Bothered very much" by blurred vision | 0
  Bothered quite a bit" or "Bothered very much" by double vision | 0
  dark area | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | The Clareon™ PanOptix™ Trifocal (Toric and Non-toric Models)
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT05518539/Prot_SAP_000.pdf